CLINICAL TRIAL: NCT02272764
Title: A Phase 1 Study of the Effects of Itraconazole on the Pharmacokinetics of ALKS 5461 in Healthy Volunteers
Brief Title: A Drug-Drug Interaction Study of ALKS 5461 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK5461-214
Record Dates: First submitted 2014-10-17; First posted 2014-10-23 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Itraconazole; ALKS 5461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Itraconazole (Other): Itraconazole or placebo
  Interventions: Drug: Itraconazole
- ALKS 5461 (Experimental): ALKS 5461 or placebo Sublingual tablet
  Interventions: Drug: ALKS 5461

INTERVENTIONS:
Drug: Itraconazole — Administered orally in a crossover design
  Other Names: Itraconazole or placebo
  Arms: Itraconazole
Drug: ALKS 5461 — Administered sublingually in a crossover design
  Other Names: ALKS 5461 or placebo
  Arms: ALKS 5461

SUMMARY:
This study will evaluate the impact of Itraconazole on the pharmacokinetics of ALKS 5461.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) of 18.0 - 30.0 kg/m2
* Is in good physical health
* Agrees to use an approved method of contraception for the duration of the study
* Additional criteria may apply

Exclusion Criteria:

* Has current evidence, or history of any clinically significant medical or psychiatric condition or observed abnormality
* Is currently pregnant or breastfeeding
* Has a history of or current infection with hepatitis B virus, hepatitis C virus, or human immunodeficiency virus (HIV)
* Has a lifetime history of opioid abuse or dependence
* Has current abuse or dependence on alcohol or any drugs
* Has used nicotine within 90 days prior to randomization
* Additional criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Drug-Drug Interaction - AUC0-t | Up to 48 hours
  Area under the concentration time curve from time zero to the last measureable time point (AUC0-t) of ALKS 5461 in the presence and absence of itraconazole
Drug-Drug Interaction - AUC0-inf | Up to 48 hours
  Area under the concentration time curve from time zero to infinity (AUC0-inf) of ALKS 5461 in the presence and absence of itraconazole
Drug-Drug Interaction - Cmax | Up to 48 hours
  Maximum plasma concentration (Cmax) of ALKS 5461 in the presence and absence of itraconazole

SECONDARY OUTCOMES:
Safety and tolerability will be measured by incidence of adverse events | Up to 32 Days

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (1):
- Alkermes Investigational Site, Overland Park, Kansas, United States